CLINICAL TRIAL: NCT00428909
Title: A Non-randomized, Open-label Study to Investigate the Effects of Imatinib Mesylate on the Pharmacokinetics of Acetaminophen/Paracetamol in Patients With Newly Diagnosed, Previously Untreated Chronic Myeloid Leukemia in Chronic Phase (CML-CP)
Brief Title: Effect of Imatinib Mesylate and the Pharmacokinetics of Acetaminophen/Paracetamol in Patients With Newly Diagnosed, Previously Untreated Chronic Myeloid Leukemia in Chronic Phase (CML-CP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571A2107
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Myeloid Leukemia (CML)
Keywords: Pharmacokinetic; STI571; imatinib; CML; Chronic Myeloid Leukemia; Philadelphia Chromosome; acetaminophen
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Philadelphia Chromosome | interventions — Imatinib Mesylate; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug-Drug interaction (Other)
  Interventions: Drug: Imatinib/Acetaminophen

INTERVENTIONS:
Drug: Imatinib/Acetaminophen

SUMMARY:
A non-randomized, open-label study to investigate the effects of imatinib mesylate on the pharmacokinetics of acetaminophen/paracetamol in patients with newly diagnosed, previously untreated chronic myeloid leukemia in chronic phase (CML-CP)

ELIGIBILITY:
Inclusion criteria:

* Ability to provide written informed consent prior to participation to the study.
* Male or female patients ≥ 18 and ≤ 75 years of age
* Patients with CML-CP within 6 months of diagnosis (date of initial diagnosis is the date of first cytogenetic analysis). FISH analysis will not be accepted.
* Diagnosis of CML in chronic phase with cytogenetic confirmation of Philadelphia chromosome of (9;22) translocations and presence of Bcr-Abl
* Documented chronic phase CML as defined by:
* < 15% blasts in peripheral blood and bone marrow
* < 30% blasts plus promyelocytes in peripheral blood and bone marrow
* < 20% basophils in the peripheral blood
* ≥ 100 x 109/L (≥ 100,000 /mm3) platelets
* No evidence of extramedullary leukemic involvement, with the exception of hepatosplenomegaly
* Adequate end organ function as defined by:
* total bilirubin < 1.5 x ULN
* SGOT and SGPT < 2.5 x UNL
* creatinine < 1.5 x ULN
* Female patients of childbearing potential must have a negative serum pregnancy test within 7 days before initiation of study drug

Exclusion criteria:

* Patients in late chronic phase, accelerated phase, or blastic phase are excluded
* Patients who have received other investigational agents
* Patients who received imatinib for any duration prior to study entry
* Patient received any treatment for CML prior to study entry for longer than 2 weeks with the exception of hydroxyurea and/or anagrelide
* Patients with another primary malignancy except if the other primary malignancy is neither currently clinically significant or requiring active intervention
* Patients who are:
* pregnant
* breast feeding
* of childbearing potential without a negative pregnancy test prior to baseline
* male or female of childbearing potential unwilling to use barrier contraceptive precautions throughout the trial
* Post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential
* Patient with a severe or uncontrolled medical condition (i.e., uncontrolled diabetes, chronic renal disease)
* Patient previously received radiotherapy to ≥ 25% of the bone marrow
* Patient had major surgery within 4 weeks prior to study entry, or who have not recovered from prior major surgery
* Patients with an ECOG Performance Status Score ≥ 3
* Patients with International normalized ratio (INR) or partial thromboplastin time (PTT) > 1.5 x IULN, with the exception of patients on treatment with oral anticoagulant
* Patients with known positivity for human immunodeficiency virus (HIV)
* baseline testing for HIV is not required
* Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent
* Patients with identified sibling donors where allogeneic bone marrow transplant is elected as first line treatment
* Patients who are chronic users of acetaminophen or medications containing acetaminophen.
* Patients who received acetaminophen or medications containing acetaminophen within 72 hours prior to study entry.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-11; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To investigate the effects of the co-administration of imatinib on the pharmacokinetics of acetaminophen / paracetamol | Day 1, day 2 -7, Day 8
To investigate the pharmacokinetic characteristics of imatinib at steady state in CML-CP patients following 400 mg dosing co-administered with acetaminophen | Day 1, Day 2-7, Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (1):
- Novartis Investigative Site, Seoul, South Korea